CLINICAL TRIAL: NCT06687070
Title: A Study of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of APG-2449 Monotherapy or in Combination With Anticancer Agents in Patients With Platinum-resistant Recurrent Ovarian Cancer or Advanced Solid Tumors
Brief Title: APG-2449 Monotherapy or in Combination With PLD in Patients With Platinum-resistant Recurrent OC or Advanced ST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG2449OC101
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Platinum-resistant Recurrent Ovarian Cancer; Advanced Solid Tumor
Keywords: APG-2449
MeSH Terms: interventions — 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APG -2449 Monotherapy (Experimental): Part A: Monotherapy for advanced solid tumors.
  Interventions: Drug: APG -2449
- APG -2449 combined with PLD (Experimental): Part B: Dose exploration and expansion of APG-2449 combined PLD.
  Interventions: Drug: APG -2449; Drug: PLD

INTERVENTIONS:
Drug: APG -2449 — Orally once a day(QD), every 28 days as a cycle.
Drug: PLD — Injected on the first day of each cycle, every 28 days as a cycle.
  Arms: APG -2449 combined with PLD

SUMMARY:
An open, multicenter, dose-exploring Phase I trial include Part A and Part B to evaluate the safety, tolerability and efficacy of APG-2449.

DETAILED DESCRIPTION:
Part A: To evaluate the safety of APG-2449 monotherapy in patients with advanced solid tumors.

Part B: To evaluate the safety, tolerability, and efficacy of APG-2449 combined with PLD in the treatment of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Part A: No gender limitation. Patients with histologically and/or cytologically confirmed ALK/ROS1 gene fusion positive non-small cell lung cancer and various advanced tumors.

   Part B: Female only. Histologically proven ovarian epithelial, fallopian tube, or primary peritoneal carcinoma.
2. At least one measurable tumor lesion.
3. ECOG score is 0~1.
4. Life expectancy of ≥3 months.
5. AE caused by previous treatment must recover to ≤ grade 1.
6. Sufficient bone marrow, liver, kidney and coagulation function.
7. Female patients must be in a non-pregnant and non-lactating state.
8. Able to understand and willing to sign informed consent.
9. Patients are required to provide fresh or archived tumor tissue samples prior to treatment.

Exclusion Criteria:

1. Undergone major surgery or major trauma within 28 days before first dose or a diagnostic biopsy within 14 days before first dose.
2. Received systemic antitumor drugs, including investigational drugs.
3. Received radiotherapy within 14 days before first dose.
4. Previous treatment with FAK inhibitors.
5. Have tumors at positions other than existing ovarian cancer or of other histological types within 3 years before first dose.
6. Known active central nervous system (CNS) metastases and/or cancerous meningitis.
7. Major cardiovascular and cerebrovascular disease occurred within 6 months before first dose.
8. Patients with pleural effusion, pericardial effusion, or ascites requiring puncture, drainage, or having received drainage within 1 month before first dose.
9. Malabsorption syndrome, or inability to take medications orally.
10. Severe gastrointestinal disease.
11. Any serious or uncontrolled systemic disease; Various chronic active infections.
12. Allergy to APG-2449 or PLD and its drug components.
13. Previous cumulative doses of anthracyclines ≥550 mg/m^2.
14. Patients using a moderately potent CYP3A4, CYP2C9, or CYP2C19 inhibitor/inducer or P-gp inhibitor within a week before first dose. Patients using CYP3A4 substrates and the drugs of a narrow treatment window within a week before first dose.
15. Other factors that, in the investigator's judgment, should prevent the patient from entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Part B: Female only.
Enrollment: 50 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events per NCI-CTCAE version 5.0. | Up to 1 year
  The number and frequency of adverse events of test drug will be assessed according to CTCAE v5.0.
Dose Limiting Toxicity(DLT). | Up to 28 days
  DLT will be defined based on the rate of drug-related grade 3 to 5 adverse events experienced within the first 4 weeks of study treatment. These will be assessed per NCI-CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jundong Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China